CLINICAL TRIAL: NCT04779125
Title: Apemesh II - Perineal Reconstruction With Mesh Enhanced Gluteus Plasty
Brief Title: APEMESH II - Perineal Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Elisa Mäkäräinen, Principal Investigator, University of Oulu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115/2020
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
Keywords: abdominoperineal resection; perineal reconstruction
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients, who have an abdominoperineal reconstruction for rectal cancer, will have a mesh enhanced gluteus plasty. The patients will be compared to historical cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluteus plasty enhanced with Progrip self gripping mesh (Experimental): All study patietns will have a gluteus enhanced plasty after abdominoperineal reconstruction.
  Interventions: Procedure: Gluteus plasty enhanced with Progrip self gripping mesh

INTERVENTIONS:
Procedure: Gluteus plasty enhanced with Progrip self gripping mesh — Intervention group will be compared to historical patients in a case-control setting. Intervention group will have a mesh enhanced gluteus plasty made to reconstruct perineum after abdominoperineal resection.

SUMMARY:
The objective of this pilot study is to assess the safety, functional outcome, feasibility and the potential benefits of synthetic mesh strip and gluteus flap reconstruction in perineum in case-control setting.

DETAILED DESCRIPTION:
Several studies have reported over 30% morbidity with perineal wound healing after abdominoperineal resection. Preoperative radiotherapy seems to be a strong predictor for perineal complications. Musculocutaneus flaps and use of biological mesh seem to minimize perineal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Curative intent abdominoperineal resection and permanent colostomy

Exclusion Criteria:

* Patient with a comorbid illness or condition that would preclude the use of surgery (ASA 4- 5)
* Immunosupression (cortisone >10mg/day) or severe malnutrition (BMI <20)
* Diabetes with 1 or more organ damage
* Dialysis treatment
* Hepatic cirrhosis Child-Bugh B-C
* Potentially curable resection not possible
* Patient undergoing emergency procedures
* Metastatic disease
* Vaginal resection, pelvic exenteration and sacrum resection
* Vaginal perforation
* Pelvic abscess or perforated tumor
* Pregnant or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Complications | 30 days
  Comprehensive complication index

SECONDARY OUTCOMES:
Surgical site infections | 30 days
  Surgical site infections
Reoperation rate | 30 days
  Reoperation rate
Operative time | 30 days
  Operative time to reconstruct perineum
Length of hospital stay | 30 days
  Primary length of stay at the hospital
Costs of treatment materials | 30 days
  Costs of treatment materials
Total perineal healing time | 1 year
  Time from operation to complete perineal healing
Perineal fistula | 30 days
  Perineal sinus or fistula
Perineal hernia | 12 months
  Perineal hernia incidence
Gluteus muscle function measured by time stands test | 12 months
  Gluteus muscle function measured by time stands test

CONTACTS AND LOCATIONS:
Overall Officials: Tero Rautio, M.D. Ph.D., Study Chair — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No